CLINICAL TRIAL: NCT03718468
Title: A Phase III, Prospective, Randomized, Open-Labeled, Active-Controlled, Multi-Center Study to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine, GC FLU, in Adults Aged 20 to 50
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT-QV-31
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC Flu Quadrivalent (Experimental)
  Interventions: Biological: GC FLU Quadrivalent
- Fluarix tetra (Active Comparator)
  Interventions: Biological: Fluarix Tetra

INTERVENTIONS:
Biological: GC FLU Quadrivalent — A single dose administration of GC FLU Quadrivalent will be through intramuscular injection.
  Arms: GC Flu Quadrivalent
Biological: Fluarix Tetra — A single dose administration of Fluarix Tetra will be through intramuscular injection.
  Arms: Fluarix tetra

SUMMARY:
This study aims to demonstrate the immunogenic efficacy of GC FLU Quadrivalent Pre-filled Syringe inj. (GC FLU), a quadrivalent influenza virus vaccine, is non-inferior to the active control, Fluarix Tetra. This study is designed to be a randomized, open-labelled, active-controlled, parallel, phase III study recruiting subjects from multiple study sites.

Approximately 840 eligible subjects are planned to enroll in order to obtain 800 evaluable (= per-protocol) subjects. Subjects will be randomized and assigned to GC FLU or Fluarix Tetra (active control, AC) group in 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Either gender, aged 20 to 50 years old (inclusive)
3. Willing and able to comply with all the required study visits and follow-up defined by this protocol
4. Female subject with childbearing potential or male subject with female spouse/partner with childbearing potential must agree to use highly effective contraceptives from 15 days prior to vaccination until 60 days after vaccination. At least two forms of birth control must be adopted and one of which must be a barrier method. Acceptable forms include:

   * Established use of oral, injected or implanted hormonal methods of contraception
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
   * Barrier methods of contraception: condom, or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Exclusion Criteria:

1. With previous known or potential exposure to influenza virus within 12 weeks prior to vaccination
2. Received seasonal influenza vaccine (registered or investigational) within 24 weeks prior to vaccination
3. Received any vaccine other than seasonal influenza vaccine within 6 weeks prior to vaccination
4. Received other investigational products (including medications and vaccines) within 6 weeks prior to vaccination
5. Administered immunoglobulins and/or other blood products within the 12 weeks prior to vaccination
6. Known or suspected hypersensitivity to any component of vaccines (including egg proteins); or history of allergy to consumption of eggs
7. History of inflammatory or degenerative neurological disease (e.g., Guillain-Barre syndrome)
8. With confirmed or suspected immunosuppressive or immunodeficient condition (e.g. HIV infection), or received > 14 days of systemic steroid with equivalent dosage equal or over to 0.5 mg/kg/day prednisolone or other immune-modifying agents within 24 weeks prior to vaccination
9. Positive in HIV, HBsAg, or HCV test
10. With fever (defined as body temperature equal or over to 38 °C by any method) on the day of vaccination
11. With ongoing acute diseases or within the past 2 years serious medical conditions (e.g. concomitant illness) such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition (e.g. alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the subject
12. Female subject who is lactating or has positive serum or urine pregnancy test at screening or vaccination

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 842 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
The Geometric Mean Titer (GMT) Ratio | 21 days after the vaccination
  The non-inferior immunogenicity of GC FLU compared to active control in terms of HAI titers against each virus strain at 21 days after the vaccination.
The Seroconversion Rate | 21 days after the vaccination
  The non-inferior immunogenicity of GC FLU compared to active control in terms of HAI titers against each virus strain at 21 days after the vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, MD, Principal Investigator — National Taiwan University Hospital
Locations (4):
- Taiwan (4):
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District